CLINICAL TRIAL: NCT00213226
Title: Efficacy of Single Dose Versus Multiple Doses of Dexamethasone in Outpatients With Acute Bronchiolitis
Brief Title: Single Dose Versus Multiple Doses of Dexamethasone in Children With Acute Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0020010349
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; pediatrics; corticosteroids
MeSH Terms: conditions — Bronchiolitis | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone

SUMMARY:
This study is to determine the effectiveness of five-day treatment versus a single dose of oral dexamethasone (corticosteroid) in children between 2 and 24 months of age with a first episode of acute bronchiolitis presenting in the Emergency Department

ELIGIBILITY:
Inclusion Criteria:

* infants 2 to 24 months of age
* acute bronchiolitis, defined as first episode of wheezing with upper respiratory infection and respiratory distress
* moderate to severe baseline disease severity (Respiratory Distress Index (RDAI) score 6 to 15)
* only patients discharged at or shortly after 240 minutes of uniform stabilization therapy will be randomized

Exclusion Criteria:

* previous wheezing and/or bronchodilator therapy
* hospitalization at 240 minutes
* critically ill patients needing airway stabilization
* patients with low or very high baseline disease severity (RDAI <5 and >16)
* patients under 8 weeks of age
* patients on corticosteroids prior to arrival at Emergency Department
* contact with varicella within 21 days
* past history of ventilation for greater than 24 hours
* existing cardiopulmonary disease, multisystem disease or immunodeficiency
* insufficient command of the English language

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2001-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients stabilized, discharged and subsequently hospitalized and/or co-interventions with corticosteroids or beta2 agonists outside the protocol within the 6 day study period

SECONDARY OUTCOMES:
Respiratory Assessment Change Score (RACS) at 96 and 144 hours
Proportion of infants with unscheduled medical visits for respiratory distress within the 6 day study period
Proportion of infants with no signs of respiratory distress at 96 and 144 hours
Proportion of infants who are symptomatic at 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Schuh S, Coates AL, Dick P, Stephens D, Lalani A, Nicota E, Mokanski M, Khaikin S, Allen U. A single versus multiple doses of dexamethasone in infants wheezing for the first time. Pediatr Pulmonol. 2008 Sep;43(9):844-50. doi: 10.1002/ppul.20845. PMID 18668692